CLINICAL TRIAL: NCT06580106
Title: A Prospective Pilot Study of the Genetic Determinants of Toxicity and Response to Azacitidine and Venetoclax in Patients With Newly Diagnosed Acute Myeloid Leukemia Through Evaluation of Polymorphisms in Pharmacokinetic Genes and Venetoclax Levels
Brief Title: Toxicity Genetic Determinants and Response to Azacitidine and Venetoclax in AML
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); Swim Across America (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00116209; LCI-LEU-AML-VENTOX-001 (Other: Atrium Health)
Record Dates: First submitted 2024-08-14; First posted 2024-08-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AML participants who are receiving or are planned to receive azacitidine plus venetoclax: Buccal swabs for SNPs and pharmacogenomic analysis can occur at any point before or after starting treatment during the study period. Venetoclax peak and trough levels will be obtained during SOC Aza/Ven treatments. CYP3A activity will also be evaluated. Demographic and cancer related history will be acquired for each participant. During study participation, cancer treatment details including administration, dose modifications, delays, and reductions, including specific grade 3 toxicities, stem cell transplant status, symptom burden, disease response, and survival will be collected. Participants will be taken off study after three years.
  Interventions: Other: Biospecimen samples

INTERVENTIONS:
Other: Biospecimen samples — Buccal swabs and Blood samples will be collected throughout study.

SUMMARY:
The purpose of this research is to see how certain genetic variations relate to side effects and outcomes experienced while receiving treatment with azacitidine and venetoclax.

DETAILED DESCRIPTION:
This is a prospective pilot study of the association of SNPs and venetoclax levels with toxicity and response to azacitidine plus venetoclax (Aza/Ven) as well as pharmacogenomics and venetoclax levels in patients with newly diagnosed AML determined to be unfit for intensive induction. Newly diagnosed AML patients over 18 years old who receive Aza/Ven as standard of care will be eligible for this study. Buccal swabs for SNPs and pharmacogenomic analysis can occur at any point before or after starting treatment during the study period. Venetoclax peak and trough levels will be obtained during SOC Aza/Ven treatments. Participants will be recruited initially at AHWFBCCC locations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.
* Age ≥ 18 years of age at the time of enrollment
* Confirmed diagnosis of AML
* Planned initial treatment with azacitidine and venetoclax
* Ability to read and understand the English and/or Spanish language
* As determined by the enrolling investigator, ability of the participant to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with AML who are receiving or are planned to receive azacitidine plus venetoclax will be identified in clinic and presented informed consent for this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity side effect | From initiation of venetoclax through 30 days after last dose
  Defined as a binary variable indicating whether a participant experienced a Grade 3 or higher of specific side effects (including infections, anemia, thrombocytopenia, febrile neutropenia, neutropenia, nausea, diarrhea)

SECONDARY OUTCOMES:
Dose Modification | Approximately 6 months or until last dose of Venetoclax, whichever came first
  A binary variable indicating whether a participant experienced a dose modification, including delay or reduction
Disease Response | Up to 3 years
  For participants diagnosed with AML, response will be defined as a binary variable indicating if they had a Complete Remission (CR), Complete Remission with partial hematologic recovery (CRh), Complete Remission with incomplete hematologic recovery (CRi), Morphologic Leukemia-free state (MLFS), or partial response (PR) to induction therapy using the European LeukemiaNet (ELN 2022) criteria. Otherwise they will be considered a non-responder
Venetoclax levels | Approx 6 months
  Will be defined as the maximum concentration of Venetoclax and is measured at 6 months if the participant is still receiving venetoclax
Overall survival | Approx 3 years
  Duration of time from date of enrollment to death. Participants who are alive or lost to follow-up at the time of the analysis will be censored at the last known date they were alive
Dose modification due to nausea or diarrhea | Approximately 6 months or until last dose of Venetoclax, whichever came first
  A binary variable indicating whether a participant experienced a dose modification, including delay or reduction due to nausea or diarrhea
Metabolizer status checklist | Approximately 6 months or until last dose of Venetoclax, whichever came first
  A categorical variable indicating whether a participant is a high, normal or low metabolizer based on pharmacogenomics analysis of SNP data

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Ragon, MD, Principal Investigator — Atrium Health Wake Forest Baptist Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No